CLINICAL TRIAL: NCT04777552
Title: The Use of Fixed-schedule Benzodiazepine Dosing Versus Treatment Based on a CIWA-Ar Alcohol Protocol in Alcohol Detoxification.
Brief Title: Fixed-schedule Benzodiazepine Dosing vs Based on a CIWA-Ar Alcohol Protocol in Alcohol Detoxification.
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Dieter Zeeuws, MD Resident Psychiatry, Universitair Ziekenhuis Brussel
Other Study IDs: 2015/298
Record Dates: First submitted 2015-12-09; First posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Alcoholdependence; CIWA-R; Benzodiazepines
MeSH Terms: interventions — Diazepam

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fixed-schedule: Untill mid 2013 patients with individually determined fixed-schedule dosage of benzodiazepines in the case of alcoholdependence.
  Interventions: Other: diazepam (or equivalence if other benzodiazepine)
- CIWA-Ar: Halfway through the year 2013 the department of psychiatry changed the protocol in alcohol withdrawal treatment and changed it to a symptom-triggered therapy with the use of CIWA-Ar to assess the severity of the alcohol withdrawal syndrome.
  Interventions: Other: diazepam (or equivalence if other benzodiazepine)

INTERVENTIONS:
Other: diazepam (or equivalence if other benzodiazepine)

SUMMARY:
Does the use of a symptom-triggered therapy (with assessment making use of a CIWA-Ar scale) decrease the total amount of benzodiazepines given to patients with alcohol dependence and are less patients still dependent on benzodiazepines on their departure in comparison with the use of a fixed-schedule dose of benzodiazepines?

DETAILED DESCRIPTION:
Methodology This study will be a retrospective study using administrative and clinical patient data of patients presenting for alcohol detoxification at the Psychiatry department of the Universitair Ziekenhuis Brussel. Two periods in the data will be compared. One period will be consisting of patient data before 2013 when the hospital still used the fixed-schedule dosing of benzodiazepines. The other period will be consisting of patient data after 2013 when the hospital switched to the symptom-triggered prescription of benzodiazepines.

Inclusion & Exclusion criteria Inclusion criteria are patients with the age of 18 years or older who were treated for alcohol .dependence at the UZ Brussel in one of the periods stated above. The criteria for exclusion were found in the literature and include pregnancy, use of central nervous system (CNS) depressant agents, history of dementia, acute psychosis, and severe hepatic dysfunction (15-18). Comorbid benzodiazepine dependence. A history of severe epilepsy on withdrawal,… Outcomes The main outcome measures will be the total amount of benzodiazepines given during the hospital stay, whether the patient is still dependent on benzodiazepines when leaving the hospital, the length of the hospital stay, and some baseline patient characteristics. These patient characteristics will include age, sex, race/ethnic group, primary reason for hospitalization, body mass index (BMI), blood alcohol level (BAL) on admission, international normalized ratio (INR), diagnosis of co-morbid psychiatric disorder, history of other substance abuse, indicators of withdrawal severity (e.g. CIWA-Ar, tremor, seizures), discharge medications, benzodiazepine dose administered (15-18).

ELIGIBILITY:
Inclusion Criteria

* patients who were treated for alcohol dependence at the UZ Brussel in one of the periods stated above.

Exclusion Criteria:

pregnancy, use of central nervous system (CNS) depressant agents, history of dementia, acute psychosis, and severe hepatic dysfunction. Comorbid benzodiazepine dependence. A history of severe epilepsy on withdrawal,…

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who were treated for alcohol dependence at the UZ Brussel in one of the periods stated above.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
total amount of benzodiazepines administrated | 7 days

IPD SHARING:
Plan to Share IPD: Undecided